CLINICAL TRIAL: NCT00027677
Title: Phase I Study To Determine The Safety Of Halofuginone In Patients With A Solid Progressive Tumor
Brief Title: Halofuginone Hydrobromide in Treating Patients With Progressive Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16007; EORTC-16007; COLLGARD-EORTC-16007
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — halofuginone

INTERVENTIONS:
Drug: halofuginone hydrobromide

SUMMARY:
RATIONALE: Halofuginone hydrobromide may stop the growth of solid tumors by stopping blood flow to the tumor.

PURPOSE: Phase I trial to study the effectiveness of halofuginone hydrobromide in treating patients who have progressive advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity profile, maximum tolerated dose, and dose-limiting toxic effects of halofuginone hydrobromide in patients with progressive advanced solid tumors.
* Establish a recommended dose of this drug for phase II study.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive oral halofuginone hydrobromide once daily on days 1 and 4-14 of course 1 and on days 1-14 of subsequent courses. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-3 patients receive escalating doses of halofuginone hydrobromide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 20% of patients experience acute dose-limiting toxicity. After the MTD is reached, 6-12 additional patients are treated at dose levels preceding the MTD until the recommended dose for phase II study is determined. The recommended dose for phase II study is defined as the dose preceding the MTD that allows a 90% dose intensity for 2 months with no greater than grade 2 toxicity in 80% of the patients.

Patients are followed every 8 weeks until disease progression or initiation of another treatment.

PROJECTED ACCRUAL: Approximately 7-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumor that is not amenable to any clinical improvement by current standard treatments

  * No tumors of the upper digestive tract
* No clinical signs of CNS involvement

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* WHO 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,000/mm^3
* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN
* No unstable hepatobiliary disease that would preclude study

Renal:

* Creatinine no greater than 1.5 times ULN
* No unstable renal disease that would preclude study

Cardiovascular:

* No unstable cardiovascular disease (e.g., stroke) that would preclude study

Pulmonary:

* No unstable pulmonary disease that would preclude study

Gastrointestinal:

* No digestive disease, including upper gastrointestinal tract, that would hamper absorption
* No evident/known lactose malabsorption

Other:

* No allergy to components of the study drug
* No uncontrolled infection
* No other unstable systemic disease that would preclude study
* No psychological, familial, sociological, or geographical condition that would preclude compliance
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior anticancer biologic therapy

Chemotherapy:

* At least 4 weeks since prior anticancer chemotherapy

Endocrine therapy:

* Prior anticancer hormonal therapy allowed

Radiotherapy:

* At least 6 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* At least 2 weeks since prior surgery

Other:

* At least 4 weeks since other prior anticancer treatment
* No other concurrent anticancer agents or investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-08; Primary Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maja De Jonge, MD, PhD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (3):
- U.Z. Gasthuisberg, Leuven, Belgium
- Netherlands (2):
  - University Hospital - Rotterdam Dijkzigt, Rotterdam
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam